CLINICAL TRIAL: NCT05501236
Title: Ansa Cervicalis and Hypoglossal Nerve Stimulation in Obstructive Sleep Apnea
Brief Title: Ansa Cervicalis and Hypoglossal Nerve Stimulation in OSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, David Kent, Assistant Professor, Department of Otolaryngology-Head and Neck Surgery, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 212305
Record Dates: First submitted 2022-07-28; First posted 2022-08-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: All patients who meet eligibility will undergo the screening sleep study, muscle stimulation during operative DISE procedure, and muscle stimulation during second sleep study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Muscle stimulation (Experimental): Consented participants who meet eligibility will have a drug induced sleep endoscopy (DISE) and second sleep study and the Grass S88 (or comparable) muscle stimulator.
  Interventions: Device: Grass S88 Muscle Stimulator

INTERVENTIONS:
Device: Grass S88 Muscle Stimulator — The Grass S88 nerve and muscle stimulator is a widely-used tool in electromyography and nerve conduction studies. During the DISE and second sleep study, fine-wire electrodes will be placed into the hypoglossal nerve or genioglossus muscle. Two more electrodes are placed transcutaneously, proximate to the bilateral branches of the cervicalis innervating the sternothyroid muscle in the anterior neck.

SUMMARY:
Polysomnography (PSG) and drug-induced sleep endoscopy (DISE) are widely used diagnostic studies for assessing obstructive sleep apnea (OSA) severity and collapse patterns of the upper airway anatomy during sleep. Hypoglossal nerve stimulation (HNS) therapy for obstructive sleep apnea suffers from variable response at the level of the soft palate. The Investigators propose a study examining the physiologic effect of ansa cervicalis stimulation (ACS) alone and in combination with HNS during PSG and DISE.

DETAILED DESCRIPTION:
Obstructive Sleep Apnea (OSA) is a common disorder characterized by repetitive upper airway collapse during inspiration caused, in part, by a loss of neuromotor tone in specific upper airway muscles, with multiple associated health sequelae impacting millions of Americans. Patient adherence to the reference treatment, positive airway pressure (PAP), remains problematic. Despite the recent promising development of hypoglossal nerve stimulation (HNS) as a surgical therapy, its indications are limited and a proportion of eligible patients do not achieve sufficient response, leaving a critical unmet need for effective therapeutic alternatives to PAP.

This project challenges the long-held concept that the genioglossus muscle is primarily responsible for the maintenance of pharyngeal patency during sleep and proposes a novel therapeutic mechanism. It is built upon strong evidence that caudal pharyngeal traction from the trachea has a marked impact on pharyngeal patency primarily mediated through changes in lung volume. Contraction of the sternothyroid muscle, an infrahyoid cervical strap muscle that inserts onto the thyroid cartilage, also generates caudal pharyngeal traction. Our data suggest that ansa cervicalis stimulation (ACS) of the sternothyroid muscle unfolds and stretches the lateral pharyngeal walls and tensions the distal edge of the soft palate caudally, increasing airway patency.

The major hypothesis of the Investigators is that ACS overcomes specific anatomic and neuromuscular defects of upper airway control that restore pharyngeal patency in patients with OSA. This hypothesis is supported by published and preliminary data demonstrating that: (1) the degree of end-expiratory lung volume decrease in sleep correlates with observed increases in pharyngeal collapsibility, and (2) unilateral ACS increases maximum inspiratory airflow and velopharyngeal cross-sectional area during flow-limited breathing in sedated humans. These findings suggest that (3) tracheal traction, as mediated by end-expiratory lung volume (EELV), is a major contributor to airway patency in sleep. In this project, the Investigators will elucidate specific mechanisms for control of pharyngeal patency with caudal traction during drug-induced sleep endoscopy (DISE) and natural sleep (PSG). The Investigators will address these aims by characterizing (1) the effects of ACS of the sternothyroid muscle(s) on upper airway pressure-area and pressure-flow relationships, and (2) determine how subject anatomic, physiologic, and polysomnographic characteristics modulate these responses.

ELIGIBILITY:
Inclusion Criteria:

1. Consenting adults with BMI≥ 25 and ≤ 40 kg/m2
2. Obstructive sleep apnea with an AHI between 20 and 80 events/hr (with hypopneas defined by 4% oxyhemoglobin desaturations); ≥80% obstructive events.

Exclusion Criteria:

1. Chronic use of opiate medications, illicit drug use, or alcohol dependency
2. Other known concomitant sleep disorder (e.g., central sleep apnea, periodic limb movements, narcolepsy)
3. Clinical history or evidence of cardiopulmonary disease (or oxygen use), liver, renal, immunodeficiency, neurodegenerative diseases, or previous adverse reactions to anesthesia.
4. Prior upper airway reconstructive surgery excluding tonsillectomy (e.g., cleft palate repair, uvulopalatopharyngoplasty)
5. Indwelling neurostimulation device (e.g. cardiac pacemaker, spinal, vagal, or hypoglossal nerve stimulator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-11-03 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Basic physiologic measurements during Drug Induced Sleep Endoscopy (DISE) - Airway cross sectional diameter | During DISE, approximately 15 minutes
  Airway cross-sectional diameter (mm^2) will be measured throughout the operative procedure via flexible fiberoptic nasopharyngoscopy.
Basic physiologic measurements during Drug Induced Sleep Endoscopy (DISE) - Airflow data | During DISE, approximately 15 minutes
  Airflow data (L/min) will be measured throughout the operative procedure via a pneumotachometer applied to the nose.
Basic physiologic measurements during Drug Induced Sleep Endoscopy (DISE) - Upper airway pressure changes | During DISE, approximately 15 minutes
  Upper airway pressure changes (cmH20) will be measured throughout the operative procedure via a pneumotachometer applied to the nose.
Basic physiologic measurements during Drug Induced Sleep Endoscopy (DISE) - Respiratory effort data | During DISE, approximately 15 minutes
  Respiratory effort data (mV) will be measured throughout the operative procedure via two respiratory inductance plethysmography belts.
Basic physiologic measurements during Polysomnography (PSG) - Airflow data | During sleep study exam (PSG), approximately 8 hours
  Airflow data (L/min) will be measured during the sleep study via a pneumotachometer applied to the nose.
Basic physiologic measurements during Polysomnography (PSG) - Electroencephalogram (EEG) | During sleep study exam (PSG), approximately 8 hours
  EEG (mV) will be collected during the sleep study via skin surface electrodes.
Basic physiologic measurements during Polysomnography (PSG) - Electrocardiogram (EKG) | During sleep study exam (PSG), approximately 8 hours
  EKG (mV) will be collected during the sleep study via skin surface electrodes.
Basic physiologic measurements during Polysomnography (PSG) - Electroocoulogram (EOG) | During sleep study exam (PSG), approximately 8 hours
  EOG (mV) will be collected during the sleep study via skin surface electrodes.
Basic physiologic measurements during Polysomnography (PSG) - Electromyography (EMG) | During sleep study exam (PSG), approximately 8 hours
  EMG data (mV) will be collected during the sleep study via skin surface electrodes.
Basic physiologic measurements during Polysomnography (PSG) - Respiratory effort data | During sleep study exam (PSG), approximately 8 hours
  Respiratory effort data (mV) will be collected during the sleep study via respiratory inductance plethysmography.
Basic physiologic measurements during Polysomnography (PSG) - Video data | During sleep study exam (PSG), approximately 8 hours
  Video data will be collected during the sleep study via in-room camera.

SECONDARY OUTCOMES:
Amount of current needed for adequate stimulation | Collected during operative and sleep study procedures, taking about 15 minutes.
  Obtain preliminary data regarding including the amount of current needed to adequately stimulate the ansa cervicalis stimulation (ACS) alone and in combination with hypoglossal nerve stimulation (HNS) during PSG and DISE via a neurostimulator connected to percutaneous electrodes.

CONTACTS AND LOCATIONS:
Overall Officials: David T. Kent, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD with other researchers.